CLINICAL TRIAL: NCT06533215
Title: Antimicrobial Efficacy of Nano-Based Intracanal Medications on Enterococcus Faecalis
Brief Title: Antimicrobial Efficacy of Nano-Based ICM on E.F
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ibrahim Ali Eissa, doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nano-Based ICM on E.F
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Enterococcus Faecalis Infection; Endodontically Treated Teeth; Endodontic Disease
Keywords: intracanal medication; Enterococcus Faecalis; secondary endodontic infection cases.
MeSH Terms: conditions — Tooth, Nonvital; Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Chlorohexidine (CHX) gel. (Active Comparator): Application of Chlorohexidine intracanal medication in secondry endodontic infection cases
  Interventions: Other: antimicrobial efficacy of nano based intracanal medications on Enterococcus faecalis count reduction in secondary endodontic infection cases.
- Group 2: Chlorohexidine loaded by silver nanoparticles (Ag-np) gel. (Active Comparator): Application of chlorohexidine loaded by silver nanoparticles (Ag-np) gel intracanal medication in secondry endodontic infection cases
  Interventions: Other: antimicrobial efficacy of nano based intracanal medications on Enterococcus faecalis count reduction in secondary endodontic infection cases.
- Group 3: Triple antibiotic-loaded chitosan nanoparticles (tachnp) gel. (Active Comparator): Application of triple antibiotic-loaded chitosan nanoparticles (tachnp) gelintracanal medication in secondry endodontic infection cases
  Interventions: Other: antimicrobial efficacy of nano based intracanal medications on Enterococcus faecalis count reduction in secondary endodontic infection cases.

INTERVENTIONS:
Other: antimicrobial efficacy of nano based intracanal medications on Enterococcus faecalis count reduction in secondary endodontic infection cases. — The paper points of three samples (S1, S2, and S3) will be placed each in a sterile falcon tube containing 1ml of brain heart infusion and labeled according to the type of intracanal medication used. Samples will be homogenized by the vortex and and one micron of each sample will be cultured on Bile Esculin Agar for E. faecalis.
  The plate will be labeled as the tube of the same sample and incubated at 37οC for 24-48 h and then after incubation, the total numbers of E.faecalis will be counted and calculated to get the colony forming units (CFU/ml).
  Other Names: Microbiological count

SUMMARY:
This in-vivo study aims to evaluate the antimicrobial effect of nano based intracanal medications (Triple antibiotic-loaded chitosan nanoparticles and chlorohexidine loaded by silver nanoparticles) on Enterococcus faecalis count reduction in secondary endodontic infection cases.

DETAILED DESCRIPTION:
Success of root canal treatment is largely dependent on the elimination of harmful microorganisms and primarily bacteria from the root canal system through chemomechanical preparation and using intracanal medication in order to cure or prevent periapical disease and allowing the maintenance of the dental element.

Failure of endodontically treated teeth is multifactorial; it is believed that the most important reason for endodontic treatment failure is the presence of microorganisms in the apical third of the root canal that survive after endodontic procedures.

Enterococcus faecalis (E. faecalis) is among the most commonly isolated bacteria from the failed endodontically treated root canals. Enterococcus is a facultative anaerobic gram-positive coccus that invades dentinal tubules, can survive in alkaline environment, endure prolonged periods of starvation, and have certain virulence factors and lytic enzymes. Its prevalence in primary endodontic infection ranges from 4% to 40 % and secondary endodontic infection ranges from 24% to 77%.

Moreover, anatomical complexity and diversity of root canals that hinders a complete disinfection of root canal space by chemo-mechanical instrumentation alone. So, the use of an intracanal medication remains an important adjunct to complete elimination of remaining bacteria by reaching areas that instruments and irrigation could not reach in addition to long-standing infections.

So, using of intracanal medication is mandatory in infected endodontic cases as more thorough debridement is achieved because of the longer overall time used for the treatment.It prevents regrowth of the remaining microbiota within the root canal system and also to increase the level of disinfection.

Chlorohexidine (CHX) is an intracanal medication that has an antibacterial effect plus high substantivity which leads to a prolonged action; however it isn't able to eradicate bacteria completely from root canals.

Triple antibiotic paste (TAP) is a combination of metronidazole, ciprofloxacin, and minocycline. This combination is able to remove diverse groups of obligate and facultative gram-positive and gram-negative bacteria, providing an environment for healing. So, this allows disinfection, and possible sterilization of the root canal system.

Introduction of nanotechnology in dentistry has been developed by using nanoparticles (NPs) exclusive features that include smaller sizes and increased surface area to volume ratio. They have higher chemical reactivity and charge density leading to greater interaction with the environment and negatively charged bacterial cells, compared to their bulk counterparts. These advantages may be used to design highly anti-microbial agents with maximal therapeutic efficacy and minimal side effects.

Intracanal medications in the nano-form can achieve optimal therapeutic activity through their interaction with microorganisms at both the sub-cellular and molecular levels. Because of their small size, they can penetrate well into the complex anatomy of the root canal system.

Chlorohexidine and triple antibiotic paste cannot be converted into nanosized forms, they can be loaded with other nanosized materials like silver and chitosan nanoparticles to gain the benefit of both materials and become nanoparticulate.

The triple antibiotic was utilized together with chitosan as a vehicle to increase its stability and controlled release of the medicament. Triple antibiotic-loaded chitosan nanoparticles (tachnp) paved the way for the use of chitosan which has an excellent antiviral, antifungal and antibacterial properties.

On the other hand, Chlorohexidine loaded by silver nanoparticles (Ag-np) had high antimicrobial efficacy which is due to the dual antibacterial effect of Ag-np and chlorohexidine, it also allowed the use of silver nanoparticles which are known for their ability to destabilize the bacterial cell membrane and increase its permeability which leads to bacterial death.

According to the current knowledge, there is limited information concerning the efficacy of different new combinations of intracanal medications on bacterial count reduction of retreatment cases. Therefore, the purpose of the present study is to evaluate the antimicrobial effect of nano-based intracanal medications on Enterococcus Faecalis in secondary endodontic infection cases.

ELIGIBILITY:
Inclusion Criteria:

* Single rooted, single canal premolar teeth.
* Teeth indicated for non-surgical root canal retreatment.
* Teeth have signs and/or symptoms of post-treatment disease manifested by recurrent acute and/or chronic periapical abscess.
* Teeth have clinical signs and symptoms of endodontic failure as sensitivity to percussion, pain, swelling or fistula.
* Teeth with radiographic features of endodontic failure as persistent periapical lesion or widening of periodontal ligament.
* Symptomatic or asymptomatic teeth with short root canal filling indicated for prosthetic restoration

Exclusion Criteria:

* Patients with any systemic diseases.
* Pregnant or lactating patients.
* Immunocompromised patients.
* Non-restorable tooth.
* Calcified root canal.
* Teeth with root fracture.
* Teeth with periodontal pocket deeper than 4mm.
* Teeth have procedural error like ledge, broken instrument, or perforation

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
the total numbers of Enterococcus Faecalis bacteria on bile esculin agar | one weak after application of intracanal medication
  colony forming units (CFU/ml).

SECONDARY OUTCOMES:
Post operative pain | one weak after application of intracanal medication
  pain on his own words

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Darrag, Phd, Principal Investigator — Professor of Endodontics; Dina Ali, phd, Study Director — Lecturer of Endodontics; Radwa Abd Elmotaleb Eissa, phd, Principal Investigator — Ass.professor of Microbiology
Locations (1):
- Faculty of Dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fahim MM, Saber SEM, Elkhatib WF, Nagy MM, Schafer E. The antibacterial effect and the incidence of post-operative pain after the application of nano-based intracanal medications during endodontic retreatment: a randomized controlled clinical trial. Clin Oral Investig. 2022 Feb;26(2):2155-2163. doi: 10.1007/s00784-021-04196-w. Epub 2021 Oct 25. PMID 34697657
- [Background] Shaik J, Garlapati R, Nagesh B, Sujana V, Jayaprakash T, Naidu S. Comparative evaluation of antimicrobial efficacy of triple antibiotic paste and calcium hydroxide using chitosan as carrier against Candida albicans and Enterococcus faecalis: An in vitro study. J Conserv Dent. 2014 Jul;17(4):335-9. doi: 10.4103/0972-0707.136444. PMID 25125845